CLINICAL TRIAL: NCT03885947
Title: Phase I Study of Valproic Acid Expanded Cord Blood Stem Cells as an Allogeneic Donor Source for Adults With Hematological Malignancies
Brief Title: VPA Expanded UCB Transplantation for Treatment of Patients With Hematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alla Keyzner (Other)
Responsible Party: Sponsor-Investigator, Alla Keyzner, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GCO 14-0451
Record Dates: First submitted 2019-03-20; First posted 2019-03-22 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Hematological Malignancy; Acute Leukemia in Remission; Acute Lymphoblastic Leukemia in Remission; Myelodysplastic Syndromes; Non-Hodgkin Lymphoma; Hodgkin Lymphoma
Keywords: Hematological Malignancies; Expanded Umbilical Cord; Allogeneic Stem Cell Transplant; Leukemia; Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia; Lymphoma | interventions — Valproic Acid; fludarabine; Cyclophosphamide; Thiotepa

STUDY DESIGN:
Intervention Model Description: Open label single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VPA expanded cord blood stem cells (Experimental): CD34 selected VPA expanded umbilical cord blood cells used in combination with or without unmanipulated umbilical cord blood for patients with hematological malignancies undergoing allogeneic stem cell transplantation.
  VPA expanded cord blood stem cells in patients with hematological malignancies undergoing allogeneic stem cell transplantation
  Interventions: Biological: Cord blood stem cells; Drug: Valproic Acid; Drug: Fludarabine; Drug: cytoxan; Drug: Thiotepa; Biological: TBI

INTERVENTIONS:
Biological: Cord blood stem cells — CD34 selected VPA expanded umbilical cord blood cells used in combination with or without unmanipulated umbilical cord blood .
Drug: Valproic Acid — Valproic Acid (VPA) expanded cord blood stem cells
  Other Names: VPA
Drug: Fludarabine — Fludarabine 150 mg/m2
Drug: cytoxan — Cytoxan 50 mg/m2
Drug: Thiotepa — Thiotepa 10 mg/m2
Biological: TBI — TBI 400cGy

SUMMARY:
In this Phase I study, the study team will evaluate the safety of Valproic Acid (VPA) expanded cord blood stem cells defined by the lack of serious infusion reactions or graft failure in patients with hematological malignancies undergoing umbilical cord blood transplantation. Moreover, the study team will also evaluate time to neutrophil and platelet engraftment as well as transplant related outcomes such as graft versus host disease (GVHD), treatment related mortality (TRM), and overall survival (OS).

DETAILED DESCRIPTION:
This is a phase I trial for safety of VPA expanded cord blood stem cells in patients with hematological malignancies undergoing allogeneic stem cell transplantation. The primary endpoint of the study is safety as defined by the incidence of infusion reactions and graft failure, lack of neutrophil engraftment by day +42. The trial will consist of two cohorts. First cohort of 5-7 patients, will undergo double umbilical cord blood (UCB) transplantation. One UCB unit will undergo CD34 selection followed VPA based expansion. CD34 negative portion of that unit will be cryopreserved to be infused later following infusion of the expanded portion. Infusion of the second unmanipulated UCB will follow it. Preparative regimen is Fludarabine 150 mg/m2/Cytoxan 50 mg/m2/Thiotepa 10 mg/m2/TBI 400cGy.

Following successful engraftment in the first cohort, second cohort (10 patients) will only receive single manipulated unit.

Otherwise, patients will receive standard allogeneic stem cell transplantation care.

ELIGIBILITY:
Inclusion Criteria:

Disease criteria:

Patients with the following hematological malignancies:

* Acute Myeloid Leukemia (AML) in complete remission (CR)
* Acute Lymphoblastic Leukemia (ALL) in complete remission (CR)
* Myelodysplastic Syndrome (MDS) requiring intensive chemotherapy
* Non-Hodgkin lymphoma in complete or partial remission
* Hodgkin lymphoma in complete or partial remission

Age Criteria:

- 18 years up to 65 years.

Organ Function and Performance Status Criteria:

- Performance status score: Karnofsky Score ≥60

Adequate major organ function defined as:

* Left ventricular ejection fraction ≥40%
* Pulmonary function test demonstrating DLCO ≥50% predicted and corrected for hemoglobin
* Serum creatinine ≤ 2 mg/dL
* Transaminases ≤ 3x ULN
* Bilirubin ≤3x ULN except for in case of Gilbert's syndrome or ongoing hemolysis
* Ability to understand and the willingness to sign a written informed consent document

Donor availability:

-Lack of suitable HLA matched related or unrelated donor available within 30 days or less if BMT is urgent in the opinion of the transplant physician.

Exclusion Criteria:

* Progressive, persistent disease or active malignancy
* Greater than 10% blasts on bone marrow biopsy in patients with MDS
* Chemotherapy naïve
* History of myelofibrosis
* Presence of Bone Marrow Fibrosis grade 2/3
* Presence of donor specific anti-HLA antibodies against available UCB units at A, B, C or DR loci, with a mean fluorescence intensity (MFI)>1000
* History of prior allogeneic stem cell transplantation
* Uncontrolled viral, bacterial or fungal infection
* History of HIV infection
* Presence of active CNS disease at the time of transplantation
* Pregnant or breastfeeding female
* Inability or unwillingness to use effective birth control.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2019-02-21 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Number of Infusion Reaction | 42 days
  Safety as measured by the incidence of infusion related reactions.
Number of Graft Failure | 42 days
  Safety as measured by the incidence of graft failures.

SECONDARY OUTCOMES:
Time to neutrophil engraftment | 1 year
  Transplant related outcomes: time to neutrophil engraftment
Time to platelets engraftment | 1 year
  Transplant related outcomes: time to platelets engraftment
Number of transplant-related mortality (TRM) | 1 year
  Transplant related outcomes: transplant-related mortality (TRM)
Number of disease free survivals | 1 year
  Transplant related outcomes: Number of disease free survivals
Number of overall survivals | 1 year
  Transplant related outcomes: Number of overall survivals
Number of participants at risk of GVHD | 1 year
  Transplant Related Outcomes: risk of GVHD
Number of infectious complications | 1 year
  Transplant Related Outcomes: incidence of infectious complications - which is any documented bacterial, viral, or fungal infections.
Time to myeloid engraftment | 42 days
  Assess the kinetics of engraftment and immune reconstitution by assessing time to myeloid engraftment
Time to lymphoid engraftment | 42 days
  Assess the kinetics of engraftment and immune reconstitution by assessing time to lymphoid engraftment
Change in T cell count | Baseline and 42 days
  Assess the kinetics of engraftment and immune reconstitution by assessing the T cell count at 42 days as compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alla Keyzner, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No